CLINICAL TRIAL: NCT04504006
Title: European Collaborative Multicenter Observational Study: Modular Treatment With PMMR and Targeted Compartmental Pelvic Lymphadenectomy Followed by Therapeutic Pelvic and Paraaortic Lymphadenectomy in Node Positive Disease for Locoregional Control in Endometrial Cancer FIGO Stages I-III
Acronym: PMMR
Status: Recruiting | Type: Observational
Sponsor: Dr. Paul Buderath (Other)
Responsible Party: Sponsor-Investigator, Dr. Paul Buderath, PD Dr. med. P. Buderath, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Other Study IDs: PMMR
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: PMMR + TCL, followed by systematic lymphadenectomy in node positive patients.
  Interventions: Procedure: Peritoneal Mesometrial Resetion + Targeted Compartmental Lymphadenectomy (PMMR+TCL)
- Cohort B: Therapy according to actual guidelines

INTERVENTIONS:
Procedure: Peritoneal Mesometrial Resetion + Targeted Compartmental Lymphadenectomy (PMMR+TCL) — Peritoneal Mesometrial Resetion + Targeted Compartmental Lymphadenectomy (PMMR+TCL)
  Groups: Cohort A

SUMMARY:
Intermediate/high risk endometrial cancer shows locoregional recurrence rates up to 20%. Also in so called low-risk disease 5-10% incidence of nodal metastasis is reported. Although adjuvant radiotherapy may reduce these recurrences there has been no survival benefit. To avoid toxicity of irradiation and preserve the full potential of radiotherapy for salvage treatment of recurrences surgery should avoid locoregional recurrence. According to the concept of ontogenetically based compartmental surgery it may be suggested that this may be achieved by PMMR and therapeutic LNE as it has been already shown for TMMR in cervical cancer and TME in rectal cancer. First, monocentric data have shown feasibility and safety of this approach and are promising with respect to reduce locoregional recurrence rate significantly. On parallel it has also been convincingly shown that sentinel node detection shows a high level of accuracy in precluding nodal involvement in endometrial cancer. Thus, unnecessary complete lymphadenectomy may be avoided in patients with proven node negative disease. However, this procedure is aimed on diagnostic and not therapeutic goals. Nevertheless, therapeutically it fits well in the surgical concept of compartmental surgery indicating the peripheral border of therapeutic surgical approach. This leads to the concept to resect the embryologically determined tissue of risk en bloc together with the "sentinel nodes" of the draining lymph compartment (module I). In case of positive node extended therapeutic pelvic and paraaortic lymphadenectomy (module II) may be indicated. This should now be evaluated in a European collaborative observational trial. The surgical arm (cohort A) will include Patients who have received surgical treatment (module I) and in case of positive nodes or enhanced risk for isolated positive paraaortic nodes (module II) and don't want to receive adjuvant radiation therapy; in intermediate/high risk situations, however, adjuvant chemotherapy should be offered to these patients. For patients with high-risk carcinomas who do not want to be treated with the modular concept, the option of receiving systematic lymphadenectomy during primary surgery will be given. Patients who prefer to be treated according current clinical practice will be asked to participate in cohort B to be observed as concomitant control and will be treated according to current clinical practice based on the European ESMO/ESGO/ESTRO-Guidelines. Primary endpoint will be loco-regional recurrence and recurrence free survival. Follow up is planned for 5 years following date of first surgery (module I).

ELIGIBILITY:
Inclusion Criteria:

* - Histologically proven endometrial carcinoma: endometroid and non-endometroid FIGO stages I-III; Karnofsky-Index ≥ 70; unrestricted operability; Age >=18 years.
* Completed treatment with according Cohort A, PMMR/targeted compartmental pelvic/paraaortic +/- complete pelvic and paraaortic LNE without adjuvant radiotherapy by the responsible clinic (clinician).

or

* Completed treatment according Cohort B, current clinical practice including adjuvant treatment based on ESMO/ESGO/ESTRO guidelines [26] by the responsible clinic (clinician).
* Informed consent of the patient

Exclusion Criteria:

* - Uterine pure sarcoma
* Distant metastases; sclerodermia, lupus erythematodes, mixed connective tissue disease; secondary malignancy; previous radiotherapy of the pelvis.
* Pregnancy
* Patients with diseases of the connective tissue will be excluded because of unforeseeable (e.g. neurological) symptoms and disorders after surgery.
* Postoperative radiotherapy could be administered with respect to the surgical field in R1 situation or if >= 5 lymph nodes were involved; in all other situations adjuvant radiotherapy will be an exclusion criterion for participation in the study cohort A. The patient may be offered documentation in analogy but apart from the study protocol.
* Patient who concomitantly participate in other studies may also be included in this study as long as inclusion criteria of this study are met, follow up data will be available and they do not experience an exclusion criterion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with the primary diagnosis of histologically proven endometrial carcinoma: endometroid and non-endometroid FIGO stages I-III; Karnofsky-Index ≥ 70; unrestricted operability; Age >=18 years.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 36 months
  Time to recurrence or progression
Intra- and postoperative complications, incidence of lymph oedema | 36 months

SECONDARY OUTCOMES:
Overall survival | 36 months
  Time to death of any cause
Rate of locoregional relapse and rate of distant metastases at 3 years. | 36 months
Pelvic organ functioning | 36 months
  Therapy-induced morbidity on bladder/urethra, rectum/bowel, vagina/vulva, assessed by the LENT-SOMA scoring system
QoL | 36 months
  Quality of life by EORTC-QLQ-C30 questionnaire at 12 and 24 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Kimmig, Prof., Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Department of Gynaecology, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No